CLINICAL TRIAL: NCT07059702
Title: Fatigue in Cerebral Palsy: An EEG- and FDG-PET-based Study of Brain Activity and Its Correlation With Fatigue.
Brief Title: Why do People With Cerebral Palsy Often Feel Fatigued?
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bjørnar Hassel, Professor, University of Oslo
Other Study IDs: REK#774384
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-07

CONDITIONS: Fatigue Intensity
Keywords: Fatigue in cerebral palsy
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with cerebral palsy: Persons with cerebral palsy of any degree, having fatigue of any degree.
  Interventions: Other: There will be no intervention.

INTERVENTIONS:
Other: There will be no intervention. — There will be no intervention. This is an observational study that uses EEG and FDG-PET results as parameters. These investigations will b e performed on a clinical basis.

SUMMARY:
Persons with cerebral palsy (CP) commonly suffer from fatigue. Fatigue is an important cause of their reduced participation in work or social life. Traditionally, CP-related fatigue has been viewed as related to the person's motor impairment. This view causes habilitation efforts to focus on muscle function. We hypothesize that the feeling of being fatigued must involve the activity of a specific, but un-identified, brain network that represents this particular sensation.

We will use electroencephalography (EEG) and 18F-2-fluoro-2-deoxyglucose positron emission tomography (FDG-PET) in CP patients with fatigue of different degrees to identify difference in brain activity that can highlight the presumed 'fatigue network' in the brain. In this work, we build on experience from another study on fatigue in people that have had a brain abscess (see: Cognitive function and fatigue after brain abscess, NCT#: NCT04938362)

Clarification of whether fatigue in CP has a muscular or cerebral cause will hopefully inform and improve habilitation efforts for this group, and it may single out fatigue as a separate treatment target.

DETAILED DESCRIPTION:
1.1. Cerebral palsy: epidemiology and symptomatology

Cerebral palsy (CP) is a neurodevelopmental disorder with a prevalence of 0.2-0.5% (Oskoui et al., 2013; McGuire et al., 2019; McIntyre et al., 2022). In most cases, the condition is apparent from early life and affects motor activity. Three phenotypes of CP are recognized according to motor disability:

spastic CP, dyskinetic CP, and atactic CP (Bekteshi et al., 2023). These variants are considered to arise from pathology affecting the corticofugal tracts, the basal ganglia, and the cerebellum, respectively.

CP is classified into 5 categories, depending on the severity of motor dysfunction (Piscitelli et al., 2021). The Gross Motor Function Classification System (GMFCS) level I means that the patient can move, walk stairs, and run and jump without any form of aid. GMFCS level II means that the patient moves with some difficulty, cannot run or jump, and need to hold a rail when walking stairs. GMFCS level III means that the patient needs a hand-held aid (stick, crutches) and needs a wheelchair for longer distances GMFCS level IV means that the patient has limited ability to move autonomously and uses a wheelchair. GMFCS level V means that the patient usually uses a wheelchair. CP has, in most cases in which a cause can be identified, a genetic background, often a de novo mutation, whereas a perinatal condition (birth asphyxia, neonatal brain infection) is a minor cause of CP (Gonzalez-Mantilla et al., 2023; Janzing et al., 2024).

1.2 Comorbidities in CP: fatigue, pain, intellectual disability, and epilepsy Fatigue is common among CP patients, affecting approximately 40% (Jacobson et al., 2020). Fatigue in CP is commonly interpreted as muscle fatigue related to the motor impairment of CP (Brunton and Rice, 2012; Puce et al., 2021). There is a growing understanding that mental fatigue is an important aspect of CP (Puce et al., 2021); however, a recent review found no valid instrument for measuring mental fatigue in CP (Dutia et al., 2024), pointing to an important obstacle in fatigue research in CP.

Pain affects approximately 50% of CP patients (van der Slot et al., 2021; Jacobson et al., 2020). Pain may originate from the musculoskeletal system related to the continuous strain on muscles, ligaments and skeleton caused by the spasticity and by the un-ergonomic postures that the patient is forced to assume during walking, in a wheelchair, or in bed. Scoliosis, hip displacement, and abdominal discomfort add to this picture. Muscle spasms, e.g., in the calves or soles of the feet, are painful, (usually) transient, muscle contractions are also common in CP (Vinkel et al., 2022). There is a strong association between pain and fatigue (Fishbain et al., 2003), which may be of particular importance in the present study.

Intellectual disability affects approximately 45% of CP patients (Reid et al., 2018). In some patients, the intellectual disability inhibits the ability to communicate the patient's need for help to alleviate their ailments, including pain (Kildal et al., 2021).

Epilepsy affects approximately 30% of CP patients (Cooper et al., 2023). As epilepsy is associated with fatigue (Kwon et al., 2017), it may contribute to the overall fatigue picture in the present study.

1.3 Fatigue in CP, a dominating symptom that is treated as a motor issue. Fatigue, together with pain, motor limitation, epilepsy, and intellectual disability, constitutes a major barrier to participation in work and social life. In our experience, fatigue is the main reason why many CP patients cannot cope in a work environment, because the constant feeling of being exhausted precludes any meaningful participation. CP is largely treated as a condition that limits motor activity. This applies to the daily or weekly physiotherapy as well as to medical treatment, such as anti-spastic treatment (botulinum toxin injections into spastic muscles and baclofen treatment) and corrective orthopedic surgery. While this treatment may also to some extent alleviate fatigue, it is our experience that CP patients continue to experience fatigue in spite of extensive treatment of motor symptoms.

1.4. A neurobiological view on fatigue: the fatigue experience is a brain phenomenon A common view is that the fatigue stems from the motor difficulties, the pain, and the spasms. However, a neurobiological view on fatigue would be that fatigue is an experience that requires a neural representation in the brain in form of a 'fatigue network'. This view lends some support from the fact that so many diseases, acute and chronic, entail fatigue, leading to the concept that many diseases and conditions can trigger this putative 'fatigue network'.

Previous work in healthy volunteers has shown that fatigue development is associated with changes in brain activity, most notably in the frontal lobes, as can be seen with electroencephalography (EEG), irrespective of the underlying cause of the fatigue (Craig et al., 2012; Perrier et al., 2016; Tran et al., 2020; Arnau et al., 2021; Pershin et al., 2023; Azadi Moghadam and Maleki, 2023). The common finding is that the band power of the alpha (8-12 Hz), theta (4-7 Hz), and delta (1-3 Hz) frequencies increases. An increase in band power reflects increased synchronous firing of neocortical neurons, which may reflect reduced frontal activity and control over other brain areas. Similar findings have been seen in fatigue-troubled patients with multiple sclerosis, cancer and fibromyalgia (Fallon et al., 2018; Keune et al., 2019; Park et al., 2019).

In some studies, fatigue has been associated with a reduction in prefrontal cerebral glucose metabolism, as can be seen with 2- 18F-2-deoxy-glucose positron emission tomography (FDG-PET). This applied to patients with multiple sclerosis(Roelcke et al., 1997) and viral hepatitis(Heeren et al., 2011).

These EEG- and FDG-PET-based studies suggest an important cerebral component in the generation of the feeling of being exhausted or fatigued.

2. Needs description There is a need to clarify whether fatigue in CP is primarily caused by muscle impairment, including peripheral musculoskeletal pain, or whether it has a predominant central nervous component. This clarification should guide habilitation efforts for this patient group, as well as enhancing the patients' understanding of themselves and their life situation.

3. Hypotheses and aims

Hypotheses:

1. We hypothesize that CP-related fatigue has an EEG- and FDG-PET signature that explains the (lack of) participation of the frontal lobes in controlling the activity of the presumed fatigue network.
2. We hypothesize that EEG and FDG-PET distinguish between severely fatigue-troubled and less severely fatigue-troubled CP patients by highlighting the activity of a presumed fatigue network.

Aims:

1. We aim to clarify whether CP-related fatigue is primarily a 'muscle phenomenon' or a 'brain phenomenon'.
2. We aim to identify the dysfunction of as yet unidentified brain areas as a main contribution to the fatigue experience in CP patients.

4. Project organization and methodology Participants are adults (>18 years old) with CP. Participants are recruited from the outpatient clinic Department of Neurohabilitation, Oslo University Hospital, where patients receive treatment with botulinum toxin and/or baclofen for spasticity on a regular basis.

EEG is performed with scalp electrodes at Oslo University Hospital. Patients are referred to the Department for Radionuclear Medicine for FDG-PET on a clinical basis to investigate the reason for their fatigue or other complaints related to their CP. We have ample experience that FDG-PET investigation of this patient group has great clinical benefit, both for correct diagnosis and for the specifics of the individual patient's everyday challenges.

4.1.2. Study design Fifty CP patients with fatigue of different degrees, from no fatigue to severely debilitating fatigue, will be included in the project. Patients will complete the Chalder's fatigue and the Fatigue severity questionnaires before undergoing EEG and FDG-PET. The Chalder's fatigue questionnaire includes an evaluation of how long the patient has experienced fatigue. 4.1.3. Risks We do not foresee major risks during the study with respect to participating patients or scientists. Under no circumstances will the study impede or delay any therapeutic interventions.

4.1.4. Statistics Patients will be allocated to one out two groups according whether their fatigue is severe or mild. CP patients with severe fatigue will be compared to patients with mild (or absence of) fatigue with respect to FDG-PET signal and EEG band power in the alpha, theta, and delta frequencies. FDG-PET results will also be compared to a normative sample that is used routinely at the Department for Radionuclear Medicine, Oslo University Hospital.

Statistical analysis will be done by parametric or non-parametric tests (1-way ANOVA or 1-way ANOVA on ranks with post-hoc tests), as appropriate. There will also be a left-right comparison of hemispheric EEG and FDG-PET data in a pairwise design.

Based on our experience with smaller sample sizes (Dahlberg 2014; 2015; 2016) we believe that a sample size of 50 CP patients is enough to discern important patterns.

4.3. Budget There is no compensation to participants or researchers in this project. Any costs are covered by the annual allowance from the University of Oslo to Professor Hassel of NOK 100 000.

4.4. Plan for activities, visibility and dissemination Results of the study will be published in peer-reviewed international medical journals. National visibility will be accomplished by publishing material on Norwegian web-based platforms.

5. User involvement The design of this study has to a large degree been conceived during clinical interviews with CP patients at The Department of Neurohabilitation, Oslo University Hospital. Their feedback (during follow-up consultations for spasticity or epilepsy treatment) will be included in the development of the study and in the interpretation of results.

6. Ethical considerations Patients with CP are frequently struggling with fatigue. While their motor impairment is often readily apparent, the fatigue is not and remains a challenge to understand for the patients themselves and for their surroundings. We feel that there is a strong ethical element in trying to disentangle the various ailments inherent in CP, and that attributing CP-related fatigue to its correct cause will enhance patients' self-understanding as well as their ability to choose wisely between habilitation alternatives. We do not see that the planned study entails serious ethical challenges for the participants, to whom their ailments are far from new; in contrast, it is our experience that CP patients find that the medical profession avoids the fatigue issue, because there is little available treatment for this aspect of CP.

7. References Arnau S, Brümmer T, Liegel N, Wascher E. Psychophysiology. 2021;58(6):e13805. doi: 10.1111/psyp.13805.

Azadi Moghadam M, Maleki A. Front Hum Neurosci. 2023;17:1248474. doi:10.3389/fnhum.2023.1248474.

Bekteshi S, Monbaliu E, McIntyre S, Saloojee G, Hilberink SR, Tatishvili N, Dan B. Towards functional improvement of motor disorders associated with cerebral palsy. Lancet Neurol. 2023;22(3):229-243. doi: 10.1016/S1474-4422(23)00004-2.

Brunton LK, Rice CL. Fatigue in cerebral palsy: a critical review. Dev Neurorehabil. 2012;15(1):54-62. doi: 10.3109/17518423.2011.629633.

Cooper MS, Mackay MT, Dagia C, Fahey MC, Howell KB, Reddihough D, Reid S, Harvey AS. Epilepsy syndromes in cerebral palsy: varied, evolving and mostly self-limited. Brain. 2023;146(2):587-599. doi: 10.1093/brain/awac274.

Craig A, Tran Y, Wijesuriya N, Nguyen H. Regional brain wave activity changes associated with fatigue. Psychophysiology. 2012;49(4):574-82. doi: 10.1111/j.1469-8986.2011.01329.x.

Dahlberg D, Ivanovic J, Hassel B. High extracellular concentration of excitatory amino acids glutamate and aspartate in human brain abscess. Neurochem Int. 2014;69:41-47.

Dahlberg D, Ivanovic J, Mariussen E, Hassel B. High extracellular levels of potassium and trace metals in human brain abscess. Neurochem Int. 2015;82:28-32.

Dahlberg D, Ivanovic J, Hassel B. Toxic levels of ammonia in human brain abscess. J Neurosurg. 2016;124:854-60 Dutia I, Eres R, Sawyer SM, Pennacchia J, Johnston LM, Cleary S, Reddihough D, Coghill D. Fatigue experienced by people with cerebral palsy: a systematic review of assessment tools and decision tree. Disabil Rehabil. 2024;46(9):1751-1759. doi: 10.1080/09638288.2023.2205175.

Fallon N, Chiu Y, Nurmikko T, Stancak A. Altered theta oscillations in resting EEG of fibromyalgia syndrome patients. Eur J Pain. 2018;22(1):49-57. doi: 10.1002/ejp.1076.

Fishbain DA, Cole B, Cutler RB, Lewis J, Rosomoff HL, Fosomoff RS. Is pain fatiguing? A structured evidence-based review. Pain Med. 2003;4(1):51-62. doi: 10.1046/j.1526-4637.2003.03008.x.

Gonzalez-Mantilla PJ, Hu Y, Myers SM, Finucane BM, Ledbetter DH, Martin CL, Moreno-De-Luca A. Diagnostic yield of exome sequencing in cerebral palsy and implications for genetic testing guidelines. JAMA Pediatr. 2023;177(5):472-478. doi:

10.1001/jamapediatrics.2023.0008. Hassel B, De Souza GA, Stensland ME, Ivanovic J, Voie Ø, Dahlberg D. The proteome of pus from human brain abscesses: host-derived neurotoxic proteins and the cell-type diversity of CNS pus. J Neurosurg. 2017;20:1-9.

Heeren M, Weissenborn K, Arvanitis D, Bokemeyer M, Goldbecker A, Tountopoulou A, Peschel T, Grosskreutz J, Hecker H, Buchert R, Berding G. J Cereb Blood Flow Metab. 2011;31(11):2199-208. doi:

10.1038/jcbfm.2011.82. Jacobson DNO, Löwing K, Tedroff K. Health-related quality of life, pain, and fatigue in young adults with cerebral palsy. Dev Med Child Neurol. 2020;62(3):372-378. doi: 10.1111/dmcn.14413.

Janzing AM, Eklund E, De Koning TJ, Eggink H. Clinical characteristics suggestive of a genetic cause in cerebral palsy: a systematic review. Pediatr Neurol. 2024;153:144-151. doi: 10.1016/j.pediatrneurol.2024.01.025.

Keune PM, Hansen S, Sauder T, Jaruszowic S, Kehm C, Keune J, Weber E, Schönenberg M, Oschmann P. Frontal brain activity and cognitive processing speed in multiple sclerosis: An exploration of EEG neurofeedback training. Neuroimage Clin. 2019;22:101716. doi: 10.1016/j.nicl.2019.101716.

Kildal E, Stadskleiv K, Boysen ES, Øderud T, Dahl IL, Seeberg TM, Guldal S, Strisland F, Morland C, Hassel B. Increased heart rate functions as a signal of acute distress in non-communicating persons with intellectual disability. Sci Rep. 2021;11(1):6479. doi: 10.1038/s41598-021-86023-6.

Kwon OY, Ahn HS, Kim HJ. Fatigue in epilepsy. Seizure. 2017;45:151-159. doi: 10.1016/j.seizure.2016.11.006.

McGuire DO, Tian LH, Yeargin-Allsopp M, Dowling NF, Christensen DL. Prevalence of cerebral palsy, intellectual disability, hearing loss, and blindness, National Health Interview Survey, 2009-2016. Disabil Health J. 2019;12(3):443-451. doi: 10.1016/j.dhjo.2019.01.005.

McIntyre S, Goldsmith S, Webb A, Ehlinger V, Hollung SJ, McConnell K, Arnaud C, Smithers-Sheedy H, Oskoui M, Khandaker G, Himmelmann K; Global CP Prevalence Group*. Global prevalence of cerebral palsy: A systematic analysis. Dev Med Child Neurol. 2022;64(12):1494-1506. doi: 10.1111/dmcn.15346.

Oskoui M, Coutinho F, Dykeman J, Jetté N, Pringsheim T. An update on the prevalence of cerebral palsy. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080.

Park HY, Jeon HJ, Bang YR, Yoon IY. Multidimensional comparison of cancer-related fatigue and chronic fatigue syndrome: the role of psychophysiological markers. Psychiatry Investig. 2019;16(1):71-79. doi: 10.30773/pi.2018.10.26.

Perrier J, Jongen S, Vuurman E, Bocca ML, Ramaekers JG, Vermeeren A. Driving performance and EEG fluctuations during on-the-road driving following sleep deprivation. Biol Psychol. 2016;121(Pt A):1-11. doi: 10.1016/j.biopsycho.2016.09.010.

Pershin I, Candrian G, Münger M, Baschera GM, Rostami M, Eich D, Müller A. Vigilance described by the time-on-task effect in EEG activity during a cued Go/NoGo task. Int J Psychophysiol. 2023;183:92-102. doi: 10.1016/j.ijpsycho.2022.11.015.

Piscitelli D, Ferrarello F, Ugolini A, Verola S, Pellicciari L. Measurement properties of the Gross Motor Function Classification System, Gross Motor Function Classification System-Expanded & Revised, Manual Ability Classification System, and Communication Function Classification System in cerebral palsy: a systematic review with meta-analysis. Dev Med Child Neurol. 2021;63(11):1251-1261. doi: 10.1111/dmcn.14910.

Puce L, Pallecchi I, Chamari K, Marinelli L, Innocenti T, Pedrini R, Mori L, Trompetto C. Systematic review of fatigue in individuals with cerebral palsy. Front Hum Neurosci. 2021;15:598800. doi: 10.3389/fnhum.2021.598800.

Reid SM, Meehan EM, Arnup SJ, Reddihough DS. Dev Med Child Neurol. 2018;60(7):687-694. doi: 10.1111/dmcn.13773.

Roelcke U, Kappos L, Lechner-Scott J, Brunnschweiler H, Huber S, Ammann W, Plohmann A, Dellas S, Maguire RP, Missimer J, Radü EW, Steck A, Leenders KL. Reduced glucose metabolism in the frontal cortex and basal ganglia of multiple sclerosis patients with fatigue: a 18F-fluorodeoxyglucose positron emission tomography study. Neurology. 1997 Jun;48(6):1566-71. doi: 10.1212/wnl.48.6.1566.

Tran Y, Craig A, Craig R, Chai R, Nguyen H. The influence of mental fatigue on brain activity: Evidence from a systematic review with meta-analyses. Psychophysiology. 2020;57(5):e13554. doi: 10.1111/psyp.13554.

van der Slot WMA, Benner JL, Brunton L, Engel JM, Gallien P, Hilberink SR, Månum G, Morgan P, Opheim A, Riquelme I, Rodby-Bousquet E, Şimşek TT, Thorpe DE, van den Berg-Emons RJG, Vogtle LK, Papageorgiou G, Roebroeck ME. Pain in adults with cerebral palsy. Ann Phys Rehabil Med. 2021;64(3):101359. doi: 10.1016/j.rehab.2019.12.011. Vinkel MN, Rackauskaite G, Finnerup NB. Classification of pain in children with cerebral palsy. Dev Med Child Neurol. 2022;64(4):447-452. doi: 10.1111/dmcn.15102

ELIGIBILITY:
Inclusion Criteria: Cerebral palsy -

Exclusion Criteria: Inability to perform EEG or FDG-PET.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with cerebral palsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG band power | From enrollment to performance of EEG at 12 weeks
  We will analyze EEG with respect to band power within alpha, theta, and delta frequencies.
  We will compare EEG results from those with mild (or absent) fatigue (a 'caseness' value of 6 or less according to Chalder's fatigue questionnaire) to those with more severe fatigue (a 'caseness' value > 6).
  We will compare EEG results from those with left-sided CP to those with right-sided CP and include those with symmetric CP (diplegic or tetraplegic CP) as reference.
EEG band power in alpha, theta, and delta frequencies | From enrollment to the performance of FDG-PET: 3 months
  FDG-PET will be analyzed with respect to regional brain activity as can be inferred from the FDG-PET signal intensity.
  We will compare FDG-PET results from those with mild/absent fatigue to those with more severe fatigue.
  We will compare FDG-PET results from those with right-sided hemiplegia to those with left-sided hemiplegia and to those with di-/tetraplegia.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurohabilitation, Oslo, Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
We do not have ethical approval to share individual data with other researchers.